CLINICAL TRIAL: NCT02863991
Title: Oral ONC201 in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to a change in corporate priorities. The decision to terminate the study was not based on any safety concerns.
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Oncoceutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC007; R01FD005402 (FDA)
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — TIC10 compound; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 375 mg ONC201 (Experimental): Patients received 375 mg ONC201 once every week in combination with dexamethasone.
  Interventions: Drug: ONC201; Drug: Dexamethasone
- 625 mg ONC201 (Experimental): Patients received 625 mg ONC201 once every week in combination with dexamethasone.
  Interventions: Drug: ONC201; Drug: Dexamethasone

INTERVENTIONS:
Drug: ONC201 — 375 mg or 625 mg ONC201
Drug: Dexamethasone — 20 mg dexamethasone

SUMMARY:
This was a Phase 1/2 open-label study of ONC201 administered orally once every week in combination with dexamethasone in adults with relapsed/refractory multiple myeloma. The primary objective of this study was to evaluate the antitumor efficacy of ONC201.

Note: This study was completed by predecessor company, Oncoceutics, Inc.

DETAILED DESCRIPTION:
In Phase 1 of the study, patients were to receive 375 or 625 mg ONC201 once every week in combination with dexamethasone using a 3+3 dose escalation design to evaluate up to 625 mg ONC201 weekly with 20 mg dexamethasone. In Phase 2 of the study, patients were to receive 625 mg ONC201 once every week. Dexamethasone was to be administered at a dose determined in Phase 1.

A treatment cycle was defined as 3 weeks. The dose-limiting toxicity window was defined as the first 3 weeks of treatment (i.e., 1 cycle). Patients may have continued treatment with ONC201 until disease progression, occurrence of an unacceptable adverse event, intercurrent illness or changes in the patient's condition rendered the patient unacceptable to continue, patient decision to withdraw from the study, or discontinuation of the study by the Sponsor.

Assessments of tumor response were conducted using the International Myeloma Working Group response criteria. Safety was assessed through the reporting of adverse events, measurement of vital signs, electrocardiograms, and clinical laboratory results.

Before the study was terminated, a total of 17 patients were enrolled and treated with ONC201: 2 patients received 375 mg ONC201 and 15 patients received 625 mg ONC201.

ELIGIBILITY:
Inclusion Criteria:

A patient had to meet all of the following criteria to be eligible to participate in the study:

1. Must have been refractory to, or not a candidate for, established therapy known to provide clinical benefit for their malignancy.
2. Had measurable disease M protein component in serum (at least 0.5 g/dL) and/or urine (if present) (≥0.2 g excreted in a 24 hour collection sample), or serum free light chain level ≥10 mg/dL, provided the serum free light chain ratio was abnormal.
3. Was able to swallow and retain oral medication.
4. Had all previous therapies for cancer, including radiotherapy, major surgery and investigational therapies discontinued for ≥14 days (≥28 days for mitomycin C or nitrosoureas) before study entry, and had all acute effects of any prior therapy resolved to baseline severity or Grade ≤1 Common Terminology Criteria for Adverse Events (CTCAE v4.03), except alopecia or parameters defined in this eligibility list.
5. Were aged ≥18 years.
6. Had an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
7. Had adequate organ and marrow function as defined below:

   1. Absolute neutrophil count: ≥1,000/mm3 without growth factor use ≤7 days prior to treatment (cycle 1 day 1, C1D1)
   2. Platelets: ≥75,000/mm3 without platelet transfusion ≤3 days prior to C1D1
   3. Hemoglobin: 8.0 mg/dL without red blood cell transfusion ≤3 days prior to C1D1
   4. Total serum bilirubin: ≤1.5 X upper limit of normal (ULN)
   5. Aspartate aminotransferase (AST) (SGOT)/alanine aminotransferase (ALT) (SGPT): ≤2 X ULN; ≤ 5 X ULN if liver dysfunction was felt to be secondary to tumor burden
   6. Serum creatinine: ≤1.5 X ULN (OR creatinine clearance ≥30 mL/min/1.73 m2)
   7. Serum or urine pregnancy test (for females of childbearing potential) negative ≤7days of starting treatment
8. Had the ability to understand and the willingness to sign a written informed consent document and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
9. Female patients must have been surgically sterile or be postmenopausal, or must have agreed to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must have been surgically sterile or must have agreed to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception was based on the judgment of the principal investigator or a designated associate.

Exclusion Criteria:

A potential patient who met any of the following criteria was ineligible to participate in the study:

1. Had active inflammatory gastrointestinal disease, chronic diarrhea (unless related to underlying malignancy or prior related treatment) or history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment. Gastroesophageal reflux disease under treatment with proton pump inhibitors was allowed.
2. Was pregnant or breast feeding.
3. Was undergoing current active treatment in another clinical study.
4. Had active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV)
5. Had known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness that was not well controlled.
6. Had active or prior plasma cell leukemia (defined as either 20% of peripheral white blood cell count [WBC] comprised of plasma/CD138+ cells or an absolute count of 2x10^9/L).
7. Had solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
8. Had serum calcium (corrected for albumin) ≥12 mg/dL
9. Had any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
10. Had other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may have increased the risk associated with study participation or study drug administration, or may have interfered with the interpretation of study results, or in the judgment of the investigator would have made the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Mount Sinai Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: 375 mg ONC201 + 20 mg Dexamethasone: Patients received 375 mg ONC201 once every week in combination with 20 mg dexamethasone.
- Phase 2: 625 mg ONC201 + 20 mg Dexamethasone: Patients received 625 mg ONC201 once every week in combination with 20 mg dexamethasone.
Period: Overall Study
Arm/Group | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone
Started | 2 | 15
Completed | 0 | 3
Not Completed | 2 | 12
Not completed — Death | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study Terminated | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: 375 mg ONC201 + 20 mg Dexamethasone: Participants received 375 mg ONC201 once weekly in combination with 20 mg dexamethasone.
- Phase 2: 625 mg ONC201 + 20 mg Dexamethasone: Participants received 625 mg ONC201 once weekly in combination with 20 mg dexamethasone.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone | Total
Number analyzed (Participants) | 2 | 15 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 11 | 12
  >=65 years | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9
  Male | 1 | 7 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 0 | 8 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 12 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Number of participants who were not a candidate for established therapy [Count of Participants; unit: Participants] — Participants with multiple myeloma and refractory and who were not a candidate for established therapy to provide clinical benefit.
  Participants | 2 | 15 | 17

OUTCOME MEASURES:

1. Primary Outcome: Response of Participants at Last On-study Visit (End of Treatment/Follow-up)
Description: Assessments of response were made using the International Myeloma Working Group (IMWG) response criteria and were assessed by magnetic resonance imaging (MRI), computed tomography (CT), or positron emission tomography (PET)/CT scans (when applicable). Per IMWG response criteria, objective response could be defined as follows: complete response (CR), disappearance of any soft tissue plasmacytomas; partial response (PR), a >50% reduction in size of soft tissue plasmacytomas; progressive disease (PD), definite development of new or a definite increase of size of existing soft tissue plasmacytomas; and stable disease (SD), not meeting criteria for CR, PR, or PD.
Time Frame: The response assessment data reported was conducted at the last on-study visit (end of treatment/follow-up), up to a maximum of 7 months following treatment initiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone
Number analyzed (Participants) | 2 | 15
Participants
  Stable disease | 1 | 2
  Progressive disease | 1 | 13

ADVERSE EVENTS:
Time Frame: From the start date and time of the first dose of study treatment up to 30 calendar days after the last dose of study treatment, up to a maximum of 7 months.
Arm/Group | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/2 | 3/15
Serious Adverse Events (participants affected / at risk) | 0/2 | 5/15
Other Adverse Events (participants affected / at risk) | 2/2 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone (N=2) | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone (N=15)
Disease progression (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Cardiac disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 375 mg ONC201 + 20 mg Dexamethasone (N=2) | Phase 2: 625 mg ONC201 + 20 mg Dexamethasone (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 13
Leukopenia (Blood and lymphatic system disorders) | 0 | 9
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8
Lacrimation increased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 11
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 4
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Swelling face (General disorders) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Carbon dioxide increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 2
Weight increased (Investigations) | 0 | 3
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6
Burning sensation (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Note: This study was terminated due to a change in corporate priorities. The decision to terminate the study was not based on any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months of the completion of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given the opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT02863991/Prot_SAP_000.pdf